CLINICAL TRIAL: NCT02617199
Title: Epidural Anesthesia as an Alternative for Management in Acute Pancreatitis, a Randomised Clinical Trial
Brief Title: Epidural Anesthesia in Acute Pancreatitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGNAE-08
Record Dates: First submitted 2015-11-14; First posted 2015-11-30 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Acute Pancreatitis
Keywords: epidural anesthesia; pain management; microcirculation
MeSH Terms: conditions — Pancreatitis; Agnosia | interventions — Anesthesia, Epidural; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural anesthesia (Experimental): Epidural anesthesia placed at L1-L2 Epidural infusion of ropivacaine 0.2% + 3-4 mcg/ml fentanyl + saline 0.9% (100 ML) 3-5ml/ hr during 120 hours
  Interventions: Drug: Epidural anesthesia
- intravenous analgesia (Active Comparator): ketorolac 1mg/kg every 8 hours or metamizol 15 mg/kg every 8 hrs and intravenous opioids (buprenorphine 3 mcg / kg or tramadol 1mg/ kg in continuos infusion
  Interventions: Drug: intravenous analgesia

INTERVENTIONS:
Drug: Epidural anesthesia — Epidural anesthesia placed at L1-L2 Epidural infusion of ropivacaine 0.2% + 3-4 mcg/ml fentanyl + saline 0.9% (100 ML) 3-5ml/ hr during 120 hours
  Other Names: ropivacaine + fentanyl epidural
  Arms: Epidural anesthesia
Drug: intravenous analgesia — ketorolac 1mg/kg every 8 hours or metamizol 15 mg/kg every 8 hrs and intravenous opioids (buprenorphine 3 mcg / kg or tramadol 1mg/ kg in continuos infusion
  Other Names: nonsteroidal analgesics + opioids intravenous
  Arms: intravenous analgesia

SUMMARY:
Acute pancreatitis is a common urgency with a mortality rate of up to 30% , decreased blood flow in the pancreatic microcirculation. It seems to be the main cause of the pathophysiology of acute pancreatitis. Today, there have been many attempts in the management of pancreatitis but no established management seems to be ideal. The epidural block is an anesthetic technique used to provide highly peri and post-operative analgesia, also plays an important role in improving the gastrointestinal vascular perfusion (due to sympathetic blockade that this technique produces) so this anesthetic technique is proposed as an alternative to both clinical treatment as an analgesic for acute pancreatitis.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the therapeutic effects of epidural block in patients with acute pancreatitis, comparing day hospital stay among patients receiving intravenous analgesic treatment and patients who are undergoing epidural block.

It is a (prospective, comparative, longitudinal, experimental, randomized) controlled clinical trial. They include patients who are diagnosed with acute pancreatitis at the Naval General Hospital of High Specialty. Two groups were taken by random assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute pancreatitis
2. Patients who agree to participate in the study

Exclusion Criteria:

1. Patients who do not agree to participate in the study
2. Patients who experience any absolute contraindication to epidural block
3. Patients with platelet counts below 80,000 mcl
4. Patients with data gastrointestinal or urinary bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Hospital days stay between two groups | 10-15 days
  Day hospital stay were compared between the analgesic management with epidural and intravenous analgesic management

SECONDARY OUTCOMES:
Efficacy of Epidural pain control | 24, 48, 72, 96,120 hours
  Measured by pain scales the effectiveness of epidural use as an analgesic in acute pancreatitis
Decreased pancreatic enzymes | 24,48,72,96,120 hours post dose
  Recording every 24 hours of laboratory values, these values decreased observing and evaluating the clinical status of the patient

OTHER OUTCOMES:
Complications associated by the epidural catheter | 24,48,72,96, 120 hours post epidural block
  Complications by epidural catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Guadalupe Ruiz Sandoval, anesthesia, Principal Investigator — Hospital General Naval de Alta Especialidad - Escuela Medico Naval
Locations (1):
- Aurora Guadalupe Ruiz Sandoval, México, D.F, Mexico City, Mexico

REFERENCES:
- [Background] Barreto SG, Saccone GT. Pancreatic nociception--revisiting the physiology and pathophysiology. Pancreatology. 2012 Mar-Apr;12(2):104-12. doi: 10.1016/j.pan.2012.02.010. Epub 2012 Feb 24. PMID 22487519
- [Result] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Result] Demirag A, Pastor CM, Morel P, Jean-Christophe C, Sielenkamper AW, Guvener N, Mai G, Berney T, Frossard JL, Buhler LH. Epidural anaesthesia restores pancreatic microcirculation and decreases the severity of acute pancreatitis. World J Gastroenterol. 2006 Feb 14;12(6):915-20. doi: 10.3748/wjg.v12.i6.915. PMID 16521220
- [Result] Steinbrook RA. Epidural anesthesia and gastrointestinal motility. Anesth Analg. 1998 Apr;86(4):837-44. doi: 10.1097/00000539-199804000-00029. No abstract available. PMID 9539611
- [Result] Hirota M, Takada T, Kitamura N, Ito T, Hirata K, Yoshida M, Mayumi T, Kataoka K, Takeda K, Sekimoto M, Hirota M, Kimura Y, Wada K, Amano H, Gabata T, Arata S, Yokoe M, Kiriyama S. Fundamental and intensive care of acute pancreatitis. J Hepatobiliary Pancreat Sci. 2010 Jan;17(1):45-52. doi: 10.1007/s00534-009-0210-7. Epub 2009 Dec 12. PMID 20012652
- [Result] Simón Hew. Acute pancreatitis: an intensive care perspective. Anteshesia and intensive care medicine. 2012; 171-175
- [Result] Frossard JL, Steer ML, Pastor CM. Acute pancreatitis. Lancet. 2008 Jan 12;371(9607):143-52. doi: 10.1016/S0140-6736(08)60107-5. PMID 18191686
- [Result] Manuel Díaz de León. Diagnóstico y tratamiento de la pancreatitis aguda grave. Medicina crítica y terapia intensiva. 2003 (17):104-10
- [Result] Skipworth JR, Pereira SP. Acute pancreatitis. Curr Opin Crit Care. 2008 Apr;14(2):172-8. doi: 10.1097/MCC.0b013e3282f6a3f9. PMID 18388680
- [Result] Siniscalchi A, Gamberini L, Laici C, Bardi T, Faenza S. Thoracic epidural anesthesia: Effects on splanchnic circulation and implications in Anesthesia and Intensive care. World J Crit Care Med. 2015 Feb 4;4(1):89-104. doi: 10.5492/wjccm.v4.i1.89. eCollection 2015 Feb 4. PMID 25685727
- [Result] J. Gil Sebrián. Analgesia y sedación en la pancreatitis aguda. Med intensiva 2003;27(2):116-28
- [Result] Layer P, Bronisch HJ, Henniges UM, Koop I, Kahl M, Dignass A, Ell C, Freitag M, Keller J. Effects of systemic administration of a local anesthetic on pain in acute pancreatitis: a randomized clinical trial. Pancreas. 2011 Jul;40(5):673-9. doi: 10.1097/MPA.0b013e318215ad38. PMID 21562445